CLINICAL TRIAL: NCT06576505
Title: Immunologiska Mekanismer Vid Sarkoidos
Brief Title: Immunological Mechanisms in Sarcoidosis
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: K2024-5925
Record Dates: First submitted 2024-08-12; First posted 2024-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sarcoidosis patients: This study only consists of one arm. The investigators follow patients prospectively and observe clinical parameters including disease course (resolving, non-resolving, which organs are involved, inflammatory markers, chest X-ray etc) and effect of treatment. In this respect the study is observational. However, the patients undergo repeated peripheral blood samples and some also undergo sampling from upper airways, faeces and a bronchoscopy and hence, the study falls in the interventional category
  Interventions: Procedure: peripheral blood sampling, bronchoscopy, upper airway and faeces sampling

INTERVENTIONS:
Procedure: peripheral blood sampling, bronchoscopy, upper airway and faeces sampling — 1. Repeated peripheral blood sampling at diagnostic and follow-up visits, in total a maximum of 400 ml/year but never more than 100 ml/ month.
  2. Upper airway sampling wih swab, aspirate and curettage, maximum 3 times/year.
  3. Faeces sampling, the patients do this themselves and leave it to the research unit, maximum 3 times/year.
  4. Bronchoscopy with lavage and a maximum of 6 mucosal biopsies before and after 6-12 months treatment.

SUMMARY:
There is no cure for the inflammatory disease sarcoidosis. Virtually any part of the body can be affected but most often the lungs and lymph nodes. Outcomes after diagnosis vary widely among sarcoidosis patients, with some experiencing resolving disease and others developing chronic disease and lung fibrosis. Cardiac sarcoidosis can lead to life threatening arrythmias and calcium metabolism disturbances can lead to renal impairment.

Treatment with different forms of immunosuppressants are usually tried to dampen symptoms but are not effective in all patients. Furthermore, the disease usually flares up after cessation of treatment. The variability in diseae course and treatment response is thought, at least to some degree, to be explained by individual differences in genetics, immune cells and signaling pathways. But existing evidence is limited. In other inflammatory diseases the gut microbiome is of importance for disease course but its role in sarcoidosis has not been clarified.

In this prospective project the investigators will study genes, inflammatory cells and signaling molecules in the lung, upper airways and blood, and to some extent microbes, also in faeces. Healthy volunteers will be included for comparative studies. Most samples will be taken during normal diagnostic work-up and follow-up of patients with/with suspected sarcoidosis. The findings will be correlated to disease course and effects of different treatments. By linking to national health data and demographic registries, comorbidities and environmental factors will be correlated to data.

By this, the investigators hope to improve understanding of which genes, cells and signaling molecules that are of importance for resolving vs non-resolving disease and why some patients respond to a certain treatment and others don´t. The overall goal is to assess and predict sarcoidosis outcomes. We hypothesize that blood-based biomarkers including those taken during routine care as well as novel cell, signaling molecules and genetic markers, in combination with clinical characteristics can be used to predict outcomes, also treatment response, in sarcoidosis. The results can lead to tailored treatment and individual follow-up for each patient with sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of sarcoidosis
* Swedish speaking
* Able to understand and approve of study protocol
* No contraindications for planned interventions
* For inclusion of healthy controls they need to be healthy and the same criteria as listed above for patients.

Exclusion Criteria:

* No suspicion of sarcoidosis
* Not Swedish-speaking
* Not able to understand study protocol
* Not approving of study protocol
* Contraindications for planned interventions

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with/with a suspicion of sarcoidosis referred to Department of Respiratory Medicine, Karolinska University Hospital, Stockholm, Sweden. A total of 4600 patients are planned to be included during 10 years (460/year).
  Healthy volunteers will be recruited through advertisments (web based platforms within Karolinska Institutet, magazines, notice-boards). A total of 400 are planned to be included during 10 years (40/year).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2024-07-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease activity | 3 months and 12 months
  This refers to cardiac sarcoidosis and is estimated with PET-CT
Number of participants with resolving vs non-resolving disease | 2 and 5 years from baseline
  Data will be collected from the medical record wether the disease resolved or not
Number of participants with immunosuppressive treatment | 5 years
  Data on treatment will be collected from the medical record
Number of participants with more than 10% change from enrollment in percent of predicted Forced Expiratory Volume in one second (L/s) at 5 years | Baseline and 5 years
  Measured with spirometry
Change from enrollment in Immunoglobulin G (g/L) at 5 years | Baseline and 5 years
  Measured in serum
Change from enrollment in fatigue at 5 years | Baseline and 5 years
  The Fatigue Assessment Scale will be used. Maximum score is 50 and minimum 10. A higher score means more fatigue.More than 22 points means the participant suffers from fatigue and more than 34 extreme fatigue.
Change from enrollment of radiographic findings at 5 years | Baseline and 5 years
  Chest X-ray will be classified according to Scadding staging
Change from enrollment of angiotensin converting enzyme (E/L) at 5 years | Baseline and 5 years
  Measured in serum
Change from enrollment of soluble Interleukin Receptor 2 (U/ml) at 5 years | Baseline and 5 years
  Measured in serum
Change from enrollment of complete blood cell count (/10x9 L) at 5 years | Baseline and 5 years
  Measured in blood
Change from enrollment of creatinine levels (micromol/L) at 5 years | Baseline and 5 years
  Measured in plasma
Change from enrollment of C-reactive protein (mg/L) at 5 years | Baseline and 5 years
  Measured in serum
Number of patients with more than 10% change from enrollment in percent of predicted Diffusing capacity of the Lungs for Carbon Monoxide (%) at 5 years | Baseline and 5 years
  Measured with spirometry
Number of participants with more than 10% change from enrollment in percent of predicted Forced Vital Capacity (L) at 5 years | Baseline and 5 years
  Measured with spirometry
Change from enrollment of calcium levels (mmol/L) at 5 years | Baseline and 5 years
  Measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: Susanna M Kullberg, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden